CLINICAL TRIAL: NCT02942706
Title: Biomarker-Panel Guided Maintenance Treatment With Cetuximab Monotherapy Versus Continuation After First Line Induction Therapy of Metastatic Colorectal Cancer (mCRC) : a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Cetuximab Maintenance Treatment Versus Continuation After Induction Therapy in mCRC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Xiangya Hospital of Central South University (Other); West China Hospital (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, MD & Ph. D, Professor of Oncology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLOC-1
Record Dates: First submitted 2016-10-02; First posted 2016-10-24 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cet maintenance (Experimental): Cetuximab maintenance treatment following induction treatment
  Interventions: Drug: Cetuximab
- Cet+chemo continuation (Active Comparator): Cetuximab plus continuation mFOLFOX6/FOLFIRI regimens
  Interventions: Drug: Cetuximab; Drug: mFOLFOX6; Drug: FOLFIRI

INTERVENTIONS:
Drug: Cetuximab — anti-EGFR monoclonal antibody
  Other Names: Erbitux
Drug: mFOLFOX6 — Oxaliplatin+LV5FU2
  Arms: Cet+chemo continuation
Drug: FOLFIRI — Irinotecan+LV5FU2
  Arms: Cet+chemo continuation

SUMMARY:
This study is try to evaluate the effect of cetuximab monotherapy as maintenance treatment, versus continuation after 8 courses of induction therapy with cetuximab plus standard chemotherapy regimen (FOLFIRI or mFOLFOX6）in metastatic colorectal cancer (mCRC) patients. The maintenance treatments are continued until disease progression or untolerated toxicity. The aim of this study is to demonstrate that cetuximab monotherapy is non-inferior to continuation treatment, in those mCRC patients who responded to induction therapy(SD, PR, or CR), and carry biomarker-panels (KRAS, NRAS, BRAF, and PIK3CA) favor EGFR antibody.

DETAILED DESCRIPTION:
This study is try to evaluate the effect of cetuximab monotherapy as maintenance treatment, versus continuation after 8 courses of induction therapy with cetuximab plus standard chemotherapy regimen (FOLFIRI or mFOLFOX6）in metastatic colorectal cancer (mCRC) patients. The maintenance treatments are continued until disease progression or untolerated toxicity. The aim of this study is to demonstrate that cetuximab monotherapy is non-inferior to continuation treatment, in those mCRC patients who responded to induction therapy(SD, PR, or CR), and carry biomarker-panels (KRAS, NRAS, BRAF, and PIK3CA) favor EGFR antibody. Furthermore, the mutation status of biomarker panel consist of KRAS, NRAS, HRAS, BRAF, EGFR, ERBB2, ERBB3, PIK3CA, PTEN, SMAD4, SMAD2, TGFBR2, cMET, Src, mTOR, VEGFR1, VEGFR2, EPHA2, MSI, TP53, ERCC1, ERCC5, KCNQ5, ILK, and Myc will be analyzed by NGS sequencing. The ctDNA as surrogate marker via liquid biopsy will be conducted before randomization, during maintenance treatment, and disease progression.

ELIGIBILITY:
Before the start of induction therapy:

Inclusion Criteria:

* Histological proof of colorectal cancer (in case of a single metastasis, histological or cytological proof of this lesion should be obtained);
* Distant metastases which are either technically unresectable or no chance to reach NED (patients with only local recurrence are not eligible);
* Measurable disease (> 1 cm on spiral CT scan or > 2 cm on chest X-ray; liver ultrasound is not allowed). Serum CEA may not be used as a parameter for disease evaluation;
* Ongoing or planned first line induction therapy with 8 cycles of FOLFIRI or mFOLFOX6.

Exclusion criteria

* Prior adjuvant treatment for stage II/III colorectal cancer ending within 6 months before the start of induction treatment
* Any prior adjuvant treatment after resection of distant metastases
* Previous systemic treatment for advanced disease
* RAS mutant mCRC

At randomisation:

Inclusion criteria:

* WHO performance status 0-1 (Karnofsky PS > 70%);
* Disease evaluation with proven SD, PR or CR according to RECIST after 8 cycles of FOLFIRI or mFOLFOX6;
* Laboratory values obtained ≤ 2 weeks prior to randomisation: adequate bone marrow function (Hb > 8.0 mmol/L, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L), renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, > 30 ml/min), liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases);
* Life expectancy > 24 weeks;
* Age: 18-75 years;
* Negative pregnancy test in women with childbearing potential;
* Expected adequacy of follow-up;
* Institutional Review Board approval;
* Written informed consent Exclusion criteria
* Chronic active infection;
* Any other concurrent severe or uncontrolled disease preventing the safe administration of study drugs;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival 1 (PFS1) | 4 months
  from randomization to progression

SECONDARY OUTCOMES:
Progression Free Survival 2 (PFS2) | 10 months
  from signing informed consent to progression
Overall Survival (OS) | 24 months
  from signing informed consent to death
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
  drug related toxicity from signing informed consent to death
Quality of life (QoL) | 24 months
  QoL from signing informed consent to death

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD & Ph.D, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wasan H, Meade AM, Adams R, Wilson R, Pugh C, Fisher D, Sydes B, Madi A, Sizer B, Lowdell C, Middleton G, Butler R, Kaplan R, Maughan T; COIN-B investigators. Intermittent chemotherapy plus either intermittent or continuous cetuximab for first-line treatment of patients with KRAS wild-type advanced colorectal cancer (COIN-B): a randomised phase 2 trial. Lancet Oncol. 2014 May;15(6):631-9. doi: 10.1016/S1470-2045(14)70106-8. Epub 2014 Apr 3. PMID 24703531
- [Background] Tveit KM, Guren T, Glimelius B, Pfeiffer P, Sorbye H, Pyrhonen S, Sigurdsson F, Kure E, Ikdahl T, Skovlund E, Fokstuen T, Hansen F, Hofsli E, Birkemeyer E, Johnsson A, Starkhammar H, Yilmaz MK, Keldsen N, Erdal AB, Dajani O, Dahl O, Christoffersen T. Phase III trial of cetuximab with continuous or intermittent fluorouracil, leucovorin, and oxaliplatin (Nordic FLOX) versus FLOX alone in first-line treatment of metastatic colorectal cancer: the NORDIC-VII study. J Clin Oncol. 2012 May 20;30(15):1755-62. doi: 10.1200/JCO.2011.38.0915. Epub 2012 Apr 2. PMID 22473155